CLINICAL TRIAL: NCT07351318
Title: Estimating Insulin Sensitivity Fluctuations Across Pregnancies With Type 1 Diabetes
Brief Title: Estimating Insulin Sensitivity in Pregnancies With Type 1 Diabetes
Acronym: EISP
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Northwestern Memorial Hospital (Other); Mount Sinai Hospital, New York (Other); Barbara Davis Center of Childhood Diabetes, University of Co (Unknown)
Responsible Party: Principal Investigator, Jacopo Pavan, Principal Investigator, University of Virginia
Other Study IDs: 20254424; 2-APF-2025-1678-A-N (Other Grant/Funding Number: BreakthroughT1D)
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Type 1 Diabetes (T1D)
Keywords: pregnancy; type 1 diabetes; diabetes; insulin; insulin sensitivity; gestation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators want to learn how the body's response to insulin changes during pregnancy in people with Type 1 Diabetes.

In this study, the investigators will look at information from people who used a Dexcom continuous glucose monitor (CGM) and a Tandem insulin pump while they were pregnant. Participants will fill out an online survey and agree to share their device data. The investigators will use this information to see how insulin sensitivity changes from three months before pregnancy to six months after the baby is born.

DETAILED DESCRIPTION:
The aim of this retrospective observational study is to collect continuous glucose monitor (CGM) and insulin pump data from pregnant individuals with Type 1 Diabetes, from 3 months before conception to 6 months after delivery. This data will be used to estimate how insulin sensitivity (IS) changes across gestation, with the goal of better understanding glucose-insulin dynamics during pregnancy and develop algorithms for adapting insulin administration across gestational ages.

Participants will complete an online survey where they will provide their insulin pump serial number, date of delivery, gestational week at delivery, date of last menstrual cycle (if known), and other optional demographic information. The study team will use this information to retrieve participants' CGM and insulin infusion data from 3 months before conception to 6 months after delivery.

Up to 200 participants will be screened, with the goal of reaching 100 screened participants.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Pregnant within the last 8 years
* Diagnosed with type 1 diabetes for at least one year at the time of pregnancy
* Use of a Dexcom CGM system (Dexcom, Inc., CA) and Tandem insulin infusion pump (Tandem Diabetes Care, CA) across gestation, and willing to share data from this pregnancy with study staff.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals with T1D who received pregnancy care within the last 8 years in one of the participating sites: UVA Health (Charlottesville, VA), Northwestern Memorial Hospital (Chicago, IL), Mount Sinai Health System (New York City, NY), Barbara Davis Center for Diabetes (Aurora, CO).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percent Time in Target Range | Assessed every 2 weeks from 4 weeks pre-conception to 6 months post partum
  Percentage of time blood glucose was 70mg/dL and 180mg/dL as per CGM

SECONDARY OUTCOMES:
Percent Time Below Range | Assessed every 2 weeks from 4 weeks pre-conception to 6 months post partum
  Percentage of time blood glucose was below 70mg/dL as per CGM
Percent Time Above Range | Assessed every 2 weeks from 4 weeks pre-conception to 6 months post partum
  Percentage of time blood glucose was above 180 mg/dl as per CGM

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Mount Sinai Hospital, New York, New York
  - UVA Health, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No